CLINICAL TRIAL: NCT07170332
Title: Clinical Study on the Safety and Efficacy of the ZIPPER™ Aortic Arch Stent-Graft System in the Treatment of Aortic Arch Dissection
Brief Title: ZIPPER™ Stent-Graft Trial for Aortic Arch Dissection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WQ202501
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Dissection of Aortic Arch
Keywords: Aortic Arch; Dissection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): The ZIPPER aortic arch stentgraft system consists of the arch mainbody stentgraft system, the branch artery stentgraft system and the thoracic extension stentgraft system.
  Interventions: Device: ZIPPER™ Stent-Graft Trial for Aortic Arch Dissection

INTERVENTIONS:
Device: ZIPPER™ Stent-Graft Trial for Aortic Arch Dissection — The ZIPPER aortic arch stentgraft system consists of the arch mainbody stentgraft system, the branch artery stentgraft system and the thoracic extension stentgraft system.

SUMMARY:
This study is the feasible study on a new technique of ZIPPER aortic arch stentgraft system

DETAILED DESCRIPTION:
The study of ZIPPER aortic arch stentgraft system is a prospective, multicenter, single arm trial, which will enroll a total of 127 patients. The goal of this study is to evaluate the safety and efficacy of ZIPPER aortic arch stentgraft system in the treatment of patients with aortic arch dissections, residual dissection following ascending aorta surgical operation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years of age.

Diagnosis and Anatomical Suitability:

Subacute or chronic aortic arch dissection requiring intervention, where the proximal end of the stent graft requires anchoring in Zone 0, and meets the following vascular anatomical criteria:

Ascending aorta (may include graft segments) ≥ 40 mm in length (measured from the sinotubular junction to the proximal edge of the IA along the centerline).

Proximal landing zone diameter ≥ 24 mm and ≤ 47 mm. Proximal landing zone length ≥ 20 mm. Diameters of the IA, LCCA, and LSA ≤ 24 mm and ≥ 6 mm, with lengths ≥ 20 mm. Suitable arterial access for endovascular intervention. Informed Consent: Capable of understanding the study purpose, voluntarily agreeing to participate, and providing written informed consent (by the subject or their legal representative). Willing to comply with follow-up requirements per the protocol.

Surgical Risk Assessment: Deemed high surgical risk (evaluated by at least two independent vascular or cardiac surgeons) or confirmed to have significant contraindications to open surgery.

Exclusion Criteria:

* Prior aortic intervention: History of open or endovascular repair of the descending or abdominal aorta.

Concurrent AAA requiring intervention: Coexisting abdominal aortic aneurysm requiring surgical intervention within 30 days.

Specific aortic pathologies: infectious aortitis, Takayasu arteritis, Marfan syndrome, or other connective tissue disorders.

Active systemic infection: Ongoing systemic infection or high risk of systemic infection.

Severe arch vessel disease: Severe stenosis, calcification, thrombosis, or tortuosity of the IA, LCCA, or LSA.

Acute ischemia: Bowel necrosis or lower limb ischemic necrosis. Pre-existing paraplegia. Post-cardiac transplant status. Recent cardiovascular events: Myocardial infarction or stroke within the past 3 months.

Advanced heart failure: NYHA Class IV or left ventricular ejection fraction (LVEF) <30%.

Active gastrointestinal bleeding: Active peptic ulcer or upper gastrointestinal bleeding within the past 3 months.

Hematologic abnormalities: Leukopenia (WBC < 3×10⁹/L), Anemia (Hb < 90 g/L), Coagulopathy, Thrombocytopenia (platelets < 50×10⁹/L).

Renal insufficiency: Serum creatinine > 221 μmol/L (2.5 mg/dL) or end-stage renal disease requiring dialysis (investigator discretion).

Severe hepatic dysfunction: ALT/AST > 5× upper limit of normal (ULN), Serum total bilirubin (STB) > 2× ULN.

High-risk intracranial lesions (any of the following):

1. Unruptured aneurysm ≥7 mm (anterior circulation) or ≥5 mm (posterior circulation)
2. Prior rupture or high-risk morphology (daughter sac, aspect ratio >1.6)
3. Intracranial arterial stenosis ≥50% with poor collateral flow. Contrast allergy. Pregnancy or lactation. Anesthesia/surgery contraindications: Severe comorbidities precluding tolerance to anesthesia or surgery.

Life expectancy < 12 months. Current participation in other drug or device clinical trials. Other exclusions: Any conditions deemed unsuitable for participation by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
30-day major adverse event (MAE)-free rate | 30 days after intervention
  Absence of the following events within 30 days post-procedure:
  All-cause mortality Ischemic stroke Myocardial infarction Renal failure: Defined as requiring persistent dialysis, renal transplantation, or leading to fatal outcomes Respiratory failure: Defined as requiring prolonged intubation (>72 hours), tracheostomy, pulmonary function deterioration, or leading to fatal outcomes Permanent paraplegia Bowel necrosis: Defined as requiring bowel resection or leading to fatal outcomes Intraoperative blood loss >1000 mL
12-month Clinical Treatment Success Rate | 12 months post-intervention
  Immediate technical success (intraoperative) Freedom from the following at 12 months post-procedure All-cause mortality. Stent graft migration (confirmed by CTA). Type I or III endoleaks (confirmed by CTA). Loss of branch stent patency (confirmed by imaging or clinical symptoms). Secondary surgical intervention

SECONDARY OUTCOMES:
All-cause mortality rate | Prior to discharge, 30 days, 6 months,12 months, 24-60 months post-procedure
Severe stroke rate (defined as modified Rankin Scale [mRS] score ≥2 at 90 days post-stroke) | Prior to discharge, 30 days, 6 months,12 months, 24-60 months post-procedure
Aortic dissection-related mortality rate | Prior to discharge, 30 days, 6 months,12 months, 24-60 months post-procedure
Major adverse event (MAE) rate | Prior to discharge, 30 days, 6 months,12 months, 24-60 months post-procedure
Device-related adverse event rate | Prior to discharge, 30 days, 6 months,12 months, 24-60 months post-procedure
Aortic dissection vascular remodeling success rate. Evaluation: Assessed via CT angiography (CTA), defined as: True lumen expansion in the stented aortic segment; False lumen reduction or obliteration; False lumen thrombosis formation. | Prior to discharge, 30 days, 6 months,12 months, 24-60 months post-procedure
Type I or III endoleak incidence rate | Prior to discharge, 30 days, 6 months,12 months, 24-60 months post-procedure
Aortic and branch stent graft migration rate | Prior to discharge, 30 days, 6 months,12 months, 24-60 months post-procedure
Postoperative branch vessel occlusion rate | Prior to discharge, 30 days, 6 months,12 months, 24-60 months post-procedure
Secondary surgical intervention rate | Prior to discharge, 30 days, 6 months,12 months, 24-60 months post-procedure

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pape LA, Awais M, Woznicki EM, Suzuki T, Trimarchi S, Evangelista A, Myrmel T, Larsen M, Harris KM, Greason K, Di Eusanio M, Bossone E, Montgomery DG, Eagle KA, Nienaber CA, Isselbacher EM, O'Gara P. Presentation, Diagnosis, and Outcomes of Acute Aortic Dissection: 17-Year Trends From the International Registry of Acute Aortic Dissection. J Am Coll Cardiol. 2015 Jul 28;66(4):350-8. doi: 10.1016/j.jacc.2015.05.029. PMID 26205591
- [Background] Evangelista A, Isselbacher EM, Bossone E, Gleason TG, Eusanio MD, Sechtem U, Ehrlich MP, Trimarchi S, Braverman AC, Myrmel T, Harris KM, Hutchinson S, O'Gara P, Suzuki T, Nienaber CA, Eagle KA; IRAD Investigators. Insights From the International Registry of Acute Aortic Dissection: A 20-Year Experience of Collaborative Clinical Research. Circulation. 2018 Apr 24;137(17):1846-1860. doi: 10.1161/CIRCULATIONAHA.117.031264. PMID 29685932